CLINICAL TRIAL: NCT04401371
Title: Comparative Evaluation of the Learning Environment of Pediatric Dentistry Course Through Hybrid Learning Versus Distance Learning
Brief Title: Distance and Hybrid Learning for Dental Student During COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Mohamed Yousry, lecturer in pediatric dentistry and dental public health, Cairo University
Other Study IDs: Distance learning environment
Record Dates: First submitted 2020-05-21; First posted 2020-05-26 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Education
Keywords: hybrid learning; distance learning; learning autonomy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hybrid learning group: students enrolled in hybrid learning pediatric dentistry course
- distance learning group: students enrolled in distance learning pediatric dentistry course

SUMMARY:
To assess dental student opinion about distance educational learning environment during COVID-19 Pandemic and to assess their satisfaction with Hybrid learning

DETAILED DESCRIPTION:
Coronavirus crisis has caused disturbance in the provision of education all over the world. In Egypt institutions of higher education has taken the decision to temporarily suspend attendance in universities and to keep it closed for student during this pandemic.

Cairo university overcome this problem by avoiding gathering and facilitating the continuity of education for all through remote learning.

In faculty of dentistry Cairo university, pediatric dentistry course coordinators and instructors made modifications in their course which is taught to 5th year dental student.

These modification included continuation of lectures and group sections through distance learning, while postponing any clinical work to avoid direct contact with patient.

In the next academic year the same course was taught in different way through hybrid learning

So the aim of the study was to compare education learning environment experiences among 5th year dental students enrolled in pediatric dentistry course through hybrid learning versus distance learning and to assess students satisfaction with hybrid learning , which will spot the light on strong and weak points in order to provide better education and improve their experiences.

ELIGIBILITY:
Inclusion Criteria:

* all 5th year dental student enrolled in pediatric dentistry hybrid and distance course in Cairo university was invited to participate

Exclusion Criteria:

* incomplete questionnaire

Ages: 20 Years to 25 Years | Sex: All
Age Groups: Adult
Study Population: 5th year dental student enrolled in pediatric dentistry hybrid and distance course in Cairo university
Sampling Method: Probability Sample
Enrollment: 376 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Comparative evaluation of education learning environment experiences among dental students enrolled in pediatric dentistry course in hybrid versus distance learning during COVID-19 crisis | 1 year
  outcome was measured by using DELES questionnaire with five items likert scale ( : 5 = always, 4 = often, 3 = sometimes, 2 = seldom, 1 = never. ranging from always to never with always representing maximum and never representing minimum always is best and never means worse questionnaire with five items likert scale ( : 5 = always, 4 = often, 3 = sometimes, 2 = seldom, 1 = never. ranging from always to never with always representing maximum and never representing minimum always is best and never means worse

SECONDARY OUTCOMES:
assessment of student satisfaction with the created environment in hybrid learning of pediatric dentistry course | 10 days
  outcome was measured by using satisfaction scale which included eight questions with answers ranging from 5 = strongly agree, 4 = agree, 3 = neither agree or disagree, 2 = disagree, 1 = strongly disagree

CONTACTS AND LOCATIONS:
Overall Officials: Yasmin Mohamed, Principal Investigator — Cairo University
Locations (1):
- Faculty of Dentistry, Cairo, Egypt

REFERENCES:
- [Derived] Yousry YM, Azab MM. Hybrid versus distance learning environment for a paediatric dentistry course and its influence on students' satisfaction: a cross-sectional study. BMC Med Educ. 2022 May 5;22(1):343. doi: 10.1186/s12909-022-03417-4. PMID 35513807